CLINICAL TRIAL: NCT03811366
Title: Multimodal Analysis and Electroretinogram in VKH From Acute Onset - a Prospective Study
Brief Title: Multimodal Analysis and Electroretinogram in VKH From Acute Onset - Part I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Joyce Hisae Yamamoto, Clinical Professor, person-in-charge of Uveitis Service, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Brazilian VKH Study Group I
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Uveomeningoencephalitic Syndrome; Inflammation; Choroid Disease; Visual Impairment
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome; Inflammation; Choroid Diseases; Vision Disorders

STUDY DESIGN:
Intervention Model Description: All patients were treated with a standard high-dose corticosteroid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Corticosteroid monotherapy (Other): All patients in the acute phase will be treated with corticosteroid monotherapy, unless presents a contraindication or persistence/ recurrence of inflammation with regressive corticosteroid monotherapy.This is the unique arm of the present study.
  Treatment protocol includes a three-day course of intravenous methylprednisolone (1000 mg per day) followed by a high dose of oral prednisone (1.0 mg/kg/day) with a slow tapering with dose equal or less than 0.1mg/kg/day after 10 months. The prednisone dose is scheduled to be reduced in a 0.1 mg/kg-step ladder until it reaches 0.3 mg/kg (i.e. for an individual with 60 kg, dose would be 20 mg): from 1 to 0.8 mg/kg every two to three weeks; at 0.7 mg/kg for 4 weeks; at 0.6 mg/kg for two to three weeks; from 0.5 mg/kg every 4 weeks; from 0.3 to 0.15 mg/kg every 6 weeks; and 0.1 mg/kg, 0.075 mg/kg and 0.05 mg/kg for 8 weeks each.
  Interventions: Drug: Corticosteroid monotherapy

INTERVENTIONS:
Drug: Corticosteroid monotherapy — Patients will receive corticosteroid monotherapy as a pulsetherapy (1000mg/ day for 3 days) followed by oral corticosteroid.
  Other Names: Prednisone arm; Corticosteroid pulsetherapy arm; Methilprednisolone arm

SUMMARY:
Patients with acute onset Vogt-Koyanagi-Harada disease (VKHD) were prospectively included in this study. They were systematically followed with clinical, posterior segment imaging exams and full-field electroretinogram during a minimum 24-month of follow-up. All patients were treated with 3-day methylprednisolone pulse therapy followed by 1mg/day oral prednisone with a slow tapper during a median of 13 months. Non-steroidal immunosuppressive therapy (IMT) was introduced in cases of refractory disease or in cases of prednisone intolerance. Outcome measured by full-field electroretinogram was analyzed and patient was grouped as electroretinogram stable or electroretinogram worsening. Clinical data was analyzed in these two electroretinogram-based groups.

DETAILED DESCRIPTION:
Consecutive patients with acute onset VKHD were included and followed for a minimum 24-month as Part I of an ongoing prospective long-term study on VKHD. The main purpose was to understand the course of clinical and subclinical choroidal inflammation in patients receiving early and high-dose corticosteroid followed by high-dose oral prednisone and a very slow tapper. All patients were followed with clinical and posterior segment imaging (PSI) exams, i.e. fundus picture, fluorescein angiography, indocyanine green angiography and enhanced depth imaging optical coherence tomography, at inclusion, 1st month, and thereof every three months. Full-field electroretinogram was performed at inclusion, 1st month, and thereof every six months. Flare was defined as appearance or increase/worsening of inflammatory signs after the initial six-month from disease onset during the predefined treatment protocol. Inflammatory signs were cells in anterior chamber, macular edema; subclinical inflammatory signs were mainly those observed by PSI exams. Scotopic full-field electroretinogram results between 12 and 24 month were the main outcome. Clinical data was analyzed in the full-field electroretinogram-based groups.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Vogt-Koyanagi-Harada disease
* acute onset with no previous treatment

Exclusion Criteria:

* non-acute VKHD
* media opacities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce H Yamamoto, PhD, Principal Investigator — Universidade São Paulo
Locations (1):
- Hospital das Clinicas HCFMUSP, Faculdade de Medicina Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Du L, Kijlstra A, Yang P. Vogt-Koyanagi-Harada disease: Novel insights into pathophysiology, diagnosis and treatment. Prog Retin Eye Res. 2016 May;52:84-111. doi: 10.1016/j.preteyeres.2016.02.002. Epub 2016 Feb 11. PMID 26875727
- [Background] Lavezzo MM, Sakata VM, Morita C, Rodriguez EE, Abdallah SF, da Silva FT, Hirata CE, Yamamoto JH. Vogt-Koyanagi-Harada disease: review of a rare autoimmune disease targeting antigens of melanocytes. Orphanet J Rare Dis. 2016 Mar 24;11:29. doi: 10.1186/s13023-016-0412-4. PMID 27008848
- [Background] Rao NA. Pathology of Vogt-Koyanagi-Harada disease. Int Ophthalmol. 2007 Apr-Jun;27(2-3):81-5. doi: 10.1007/s10792-006-9029-2. Epub 2007 Apr 14. PMID 17435969
- [Background] Rubsamen PE, Gass JD. Vogt-Koyanagi-Harada syndrome. Clinical course, therapy, and long-term visual outcome. Arch Ophthalmol. 1991 May;109(5):682-7. doi: 10.1001/archopht.1991.01080050096037. PMID 2025171
- [Background] Herbort CP Jr, Abu El Asrar AM, Takeuchi M, Pavesio CE, Couto C, Hedayatfar A, Maruyama K, Rao X, Silpa-Archa S, Somkijrungroj T. Catching the therapeutic window of opportunity in early initial-onset Vogt-Koyanagi-Harada uveitis can cure the disease. Int Ophthalmol. 2019 Jun;39(6):1419-1425. doi: 10.1007/s10792-018-0949-4. Epub 2018 Jun 11. PMID 29948499
- [Background] Yang P, Fang W, Wang L, Wen F, Wu W, Kijlstra A. Study of macular function by multifocal electroretinography in patients with Vogt-Koyanagi-Harada syndrome. Am J Ophthalmol. 2008 Nov;146(5):767-71. doi: 10.1016/j.ajo.2008.05.044. Epub 2008 Jul 30. PMID 18672226
- [Background] Chee SP, Jap A, Bacsal K. Spectrum of Vogt-Koyanagi-Harada disease in Singapore. Int Ophthalmol. 2007 Apr-Jun;27(2-3):137-42. doi: 10.1007/s10792-006-9009-6. Epub 2006 Nov 11. PMID 17103022
- [Background] Yuan W, Zhou C, Cao Q, Du Z, Hu R, Wang Y, Kijlstra A, Yang P. Longitudinal Study of Visual Function in Vogt-Koyanagi-Harada Disease Using Full-Field Electroretinography. Am J Ophthalmol. 2018 Jul;191:92-99. doi: 10.1016/j.ajo.2018.04.013. Epub 2018 Apr 25. PMID 29702075
- [Background] Chee SP, Luu CD, Cheng CL, Lim WK, Jap A. Visual function in Vogt-Koyanagi-Harada patients. Graefes Arch Clin Exp Ophthalmol. 2005 Aug;243(8):785-90. doi: 10.1007/s00417-005-1156-3. Epub 2005 Mar 11. PMID 15761760
- [Background] da Silva FT, Hirata CE, Olivalves E, Oyamada MK, Yamamoto JH. Fundus-based and electroretinographic strategies for stratification of late-stage Vogt-Koyanagi-Harada disease patients. Am J Ophthalmol. 2009 Dec;148(6):939-45.e3. doi: 10.1016/j.ajo.2009.06.029. Epub 2009 Sep 24. PMID 19781687
- [Background] Tugal-Tutkun I, Herbort CP, Khairallah M; Angiography Scoring for Uveitis Working Group (ASUWOG). Scoring of dual fluorescein and ICG inflammatory angiographic signs for the grading of posterior segment inflammation (dual fluorescein and ICG angiographic scoring system for uveitis). Int Ophthalmol. 2010 Oct;30(5):539-52. doi: 10.1007/s10792-008-9263-x. Epub 2008 Sep 16. PMID 18795232
- [Background] Nakayama M, Keino H, Watanabe T, Okada AA. Clinical features and visual outcomes of 111 patients with new-onset acute Vogt-Koyanagi-Harada disease treated with pulse intravenous corticosteroids. Br J Ophthalmol. 2019 Feb;103(2):274-278. doi: 10.1136/bjophthalmol-2017-311691. Epub 2018 Apr 17. PMID 29666121
- [Background] Kawaguchi T, Horie S, Bouchenaki N, Ohno-Matsui K, Mochizuki M, Herbort CP. Suboptimal therapy controls clinically apparent disease but not subclinical progression of Vogt-Koyanagi-Harada disease. Int Ophthalmol. 2010 Feb;30(1):41-50. doi: 10.1007/s10792-008-9288-1. Epub 2009 Jan 17. PMID 19151926
- [Background] Herbort CP Jr, Abu El Asrar AM, Yamamoto JH, Pavesio CE, Gupta V, Khairallah M, Tugal-Tutkun I, Soheilian M, Takeuchi M, Papadia M. Reappraisal of the management of Vogt-Koyanagi-Harada disease: sunset glow fundus is no more a fatality. Int Ophthalmol. 2017 Dec;37(6):1383-1395. doi: 10.1007/s10792-016-0395-0. Epub 2016 Nov 14. PMID 27844182
- [Background] Abu El-Asrar AM, Dosari M, Hemachandran S, Gikandi PW, Al-Muammar A. Mycophenolate mofetil combined with systemic corticosteroids prevents progression to chronic recurrent inflammation and development of 'sunset glow fundus' in initial-onset acute uveitis associated with Vogt-Koyanagi-Harada disease. Acta Ophthalmol. 2017 Feb;95(1):85-90. doi: 10.1111/aos.13189. Epub 2016 Aug 18. PMID 27535102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment: June, 2011 through January, 2017 Location: Ophthalmology service -Hospital das Clínicas da Universidade São Paulo
Units Other Than Participants: Eyes
Groups:
- Corticosteroid Monotherapy: All patients in the acute phase will be treated with corticosteroid monotherapy, unless presents a contraindication or persistence/ recurrence of inflammation with regressive corticosteroid monotherapy.
  Treatment protocol includes a three-day course of intravenous methylprednisolone (1000 mg per day) followed by a high dose of oral prednisone (1.0 mg/kg/day) with a slow tapering with dose equal or less than 0.1mg/kg/day after 10 months. The prednisone dose is scheduled to be reduced in a 0.1 mg/kg-step ladder until it reaches 0.3 mg/kg (i.e. for an individual with 60 kg, dose would be 20 mg): from 1 to 0.8 mg/kg every two to three weeks; at 0.7 mg/kg for 4 weeks; at 0.6 mg/kg for two to three weeks; from 0.5 mg/kg every 4 weeks; from 0.3 to 0.15 mg/kg every 6 weeks; and 0.1 mg/kg, 0.075 mg/kg and 0.05 mg/kg for 8 weeks each.
Period: Overall Study
Arm/Group | Corticosteroid Monotherapy
Started | 12; 24 Eyes
Completed | 12; 24 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Study of clinical, subclinical and electroretinographic outcomes of patients with acute Vogt-Koyanagi-Harada disease treated with corticosteroid monotherapy
Groups:
- Corticosteroid Monotherapy: All patients in the acute phase will be treated with corticosteroid monotherapy, unless presents a contraindication or persistence/ recurrence of inflammation with regressive corticosteroid monotherapy.
  Treatment protocol includes a three-day course of intravenous methylprednisolone (1000 mg per day) followed by a high dose of oral prednisone (1.0 mg/kg/day) with a slow tapering with dose equal or less than 0.1mg/kg/day after 10 months. The prednisone dose is scheduled to be reduced in a 0.1 mg/kg-step ladder until it reaches 0.3 mg/kg (i.e. for an individual with 60 kg, dose would be 20 mg): from 1 to 0.8 mg/kg every two to three weeks; at 0.7 mg/kg for 4 weeks; at 0.6 mg/kg for two to three weeks; from 0.5 mg/kg every 4 weeks; from 0.3 to 0.15 mg/kg every 6 weeks; and 0.1 mg/kg, 0.075 mg/kg and 0.05 mg/kg for 8 weeks each.
  prednisolone and prednisone
Arm/Group | Corticosteroid Monotherapy
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 31 [15 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 12

OUTCOME MEASURES:

1. Primary Outcome: Median Values of ERG Scotopic Parameters at 12-month
Description: Full-field electroretinogram (ERG) scotopic parameters were evaluated at 12 -month (scotopic parameters: amplitude of scotopic a and b wave, amplitude of maximum scotopic a and b wave, oscillatory potential).
Time Frame: assessed at 12-month
Measure: Median (Full Range); unit: microvolts
Units Other Than Participants: eyes
Arm/Group | Corticosteroid Monotherapy
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
microvolts
  Scotopic b amplitude | 201 [104 to 352]
  Maximum scotopic a amplitude | 210 [134 to 336]
  Maximum scotopic b amplitude | 508 [328 to 728]
  Oscillatory potential | 92 [48 to 272]
  Photopic a amplitude | 42 [23 to 63]
  Photopic B amplitude | 202 [87 to 312]
  Flicker | 52 [24 to 89]
Statistical Analysis 1: Comparison: Corticosteroid Monotherapy; Test type: Other; p < 0.001, generalized estimated equation — significance when p<0;05; generalized estimated equation with normal distribution and logarithmic link function

2. Primary Outcome: Median Values of ERG Scotopic Parameters at 24-month
Description: Full-field electroretinogram (ERG) scotopic parameters were evaluated at 24 -month (scotopic parameters: amplitude of scotopic a and b wave, amplitude of maximum scotopic a and b wave, oscillatory potential).
Time Frame: assessed at 24-month
Measure: Median (Full Range); unit: microvolts
Units Other Than Participants: eyes
Arm/Group | Corticosteroid Monotherapy
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
microvolts
  Scotopic b amplitude | 189 [130 to 380]
  Maximum scotopic a amplitude | 189 [120 to 317]
  Maximum scotopic b amplitude | 484 [336 to 789]
  Oscillatory potential | 114 [35 to 259]
  Photopic a amplitude | 43 [23 to 66]
  Photopic B amplitude | 186 [111 to 345]
  Flicker | 54 [29 to 85]

3. Primary Outcome: Variation (Worsening or Improvement) Between 24 and 12 Months of ERG Scotopic Parameters Comparing 24 and 12-months
Description: Full-field electroretinogram (ERG) scotopic parameters at 12 and 24 months were compared (scotopic parameters: amplitude of scotopic a and b wave, amplitude of maximum scotopic a and b wave, oscillatory potential). The worsening of the ERG parameters was defined as a value reduction of ≥ 30 % in any these scotopic ERG parameters at month 12 and month 24. We report the change between the (value at month 24/ the value at month 12)*100.
Time Frame: 12 and 24-months
Population: One patient had an eye classified as ERG stable group and the other eye as ERG worsening group thus the sum of both groups exceed the total 12 participants
Measure: Number; unit: percentage of change on ERG parameters
Units Other Than Participants: eyes
Groups:
- ERG Stable Group: The stability of the ERG parameters was defined as a value reduction of < 30 % in any scotopic ERG parameter, which was confirmed in two consecutive examinations
- ERG Worsening Group: The worsening of the ERG parameters was defined as a value reduction of ≥ 30 % in any scotopic ERG parameter, which was confirmed in two consecutive examinations
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
percentage of change on ERG parameters
  Scotopic b amplitude | 9.5 | -32.9
  Maximum scotopic a amplitude | 7 | -21.4
  Maximum scotopic b amplitude | 2.8 | -10.8
  Oscillatory potential | 5.9 | -47.1
  Photopic a amplitude | 0 | -5
  Photopic b amplitude | 2.4 | -13.6
  Flicker | 6.2 | -6.9

4. Secondary Outcome: Recurrence or Worsening of Cells in Anterior Chamber
Description: Evaluation of anterior chamber (AC) cells was performed at visits 6 months, 12 months, 18 months and 24 months from disease onset, according to the Standardization of Uveitis Nomenclature´s classification of anterior chamber cells. (Am J Ophthalmol, 2005) Any step increase (fluctuation), when comparing sequential dates of follow up (e.g 6 and 12 months) were considered as one episode of clinical worsening in AC cells
Time Frame: 6 to 24 months from disease onset.
Population: as for outcome 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 8 | 0
Statistical Analysis 1: Comparison: ERG Stable Group vs ERG Worsening Group; Recurrence or worsening of cells in anterior chamber in ERG-stable and ERG worsening group; Test type: Other; p = 0.054, Fisher Exact — significance when p<0.05

5. Secondary Outcome: Increase in the Score of Dark Dots on Indocyanine Green Angiography
Description: Dark dots scores had a maximum value of 8, any increase of 0.5 after 6 months from disease onset will be considered (Int Ophthalmo 2010) Dark dots Score based on pattern of distribution (Sparse/ Numerous) Minimum: 0 (better outcome) Maximum: 8 (worse outcome)
Time Frame: 6 to 24 months from disease onset
Population: as for outcome 3
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- ERG Worsening-group: The worsening of the ERG parameters was defined as a value reduction of ≥ 30 % in any scotopic ERG parameter, which was confirmed in two consecutive examinations
Arm/Group | ERG Stable Group | ERG Worsening-group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 17 | 5
Statistical Analysis 1: Comparison: ERG Stable Group; Test type: Other; p = 0.478, generalized estimated equation — 17 eyes presented dark dots fluctuation during follow up in stable ERG group when compared to 5 eyes in worsening ERG group; Generalized estimated equation with Poisson distribution and identity link function supposing an interchangeable correlation matrix between the eyes

6. Secondary Outcome: Change in Subfoveal Choroidal Thickness on Enhanced Depth Optical Coherence Tomography
Description: Increase of 30% or more in choroidal thickness EDI in consecutive exams on horizontal scan
Time Frame: 6 to 24 months from disease onset
Population: as for outcome 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- ERG Worsening-group: he worsening of the ERG parameters was defined as a value reduction of ≥ 30 % in any scotopic ERG parameter, which was confirmed in two consecutive examinations
Arm/Group | ERG Stable Group | ERG Worsening-group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 8 | 4

7. Secondary Outcome: Change in Perivascular Leakage on Fluorescein Angiography
Description: Perivascular leakage was observed as an increase in hyperfluorescence around retinal vasculature over time on FA exam at midperiphery.
Time Frame: 6 to 24 months after disease onset
Population: as for outcome 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 9 | 4
Statistical Analysis 1: Comparison: ERG Stable Group; Change in perivascular leakage in ERG-stable and ERG- worsening groups; Test type: Other — 9 (52.9%) eyes in ERG stable group x 4 (57.1%)eyes presented change in perivascular leakage during follow up (p=0.936); p = 0.936, Generalized estimated equation; Generalized estimated equation with binomial distribution and logit link function, supposing an interchangeable correlation matrix between the eyes;

8. Secondary Outcome: Choroidal Neovascularization
Description: Choroidal neovascularization was diagnosed when increasingly localized hyperfluorescence at the posterior pole is detected on FA or a hyperreflective subretinal lesion associated with sub or intraretinal fluid on OCT.
Time Frame: 6 to 24 months after disease onset
Population: as for outcome 3
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 2 | 1
Statistical Analysis 1: Comparison: ERG Stable Group vs ERG Worsening Group; Test type: Other; p = 0.853, Generalized estimated equation — significance when p<0.05; [statistical method as in outcome 7, analysis 1]

9. Secondary Outcome: Cataract
Description: Cataract was defined as any lens opacification greater than nuclear or cortical 2+/4 or subcapsular 1+/4
Time Frame: 6 to 24 months after disease onset
Population: as for outcome 3
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 5 | 0
Statistical Analysis 1: Comparison: ERG Stable Group vs ERG Worsening Group; Test type: Other; p = 0.272, Fisher Exact — significance when p<0.05

10. Secondary Outcome: Ocular Hypertension
Description: Ocular hypertension was defined as an intraocular pressure (IOP) above 21mmHg
Time Frame: 6 to 24 months after disease onset
Population: as for outcome 3
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | ERG Stable Group | ERG Worsening Group
Number analyzed (Participants) | 9 | 4
Number analyzed (eyes) | 17 | 7
eyes | 7 | 5
Statistical Analysis 1: Comparison: ERG Stable Group vs ERG Worsening Group; Test type: Other; p = 0.983, Generalized estimated equation with bino — significance when p<0.05; Generalized estimated equation with binomial distribution and logit link function, supposing an interchangeable correlation matrix between the eyes

ADVERSE EVENTS:
Time Frame: 12 and 24 months
Description: 1. Weight gain
  2. Psychosis/ Depression
Arm/Group | Corticosteroid Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid Monotherapy (N=12)
Psychosis/ depression (Psychiatric disorders) | 2 (2) — Psychosis/ depression
Weight gain (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT03811366/Prot_SAP_002.pdf
  • Informed Consent Form (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT03811366/ICF_003.pdf